CLINICAL TRIAL: NCT00408265
Title: Smoking Cessation in Substance Abuse Treatment Patients: A Feasibility Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAA-ALE-03510; NIH Grant P50-AA03510
Record Dates: First submitted 2006-12-04; First posted 2006-12-06 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Nicotine Dependence
Keywords: Nicotine Dependence; Contingency Management
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Contingency Management

SUMMARY:
The purpose of this study is to compare the effects of self-help materials for smoking cessation and self-help materials for smoking cessation plus prize-based contingency management (CM), in which prize incentives are available for breath and saliva samples that indicate smoking abstinence, in substance abuse treatment patients who want to quit smoking.

DETAILED DESCRIPTION:
The specific aims of this study are: (1) to examine the efficacy of self-help materials compared to self-help materials plus prize contingency management (CM) for smoking abstinence in substance abuse treatment patients and (2) examine the effects of smoking abstinence on substance use and substance treatment retention. To address these specific aims, cigarette smokers entering treatment for alcohol, cocaine or heroin abuse or dependence, who report daily smoking (at least one cigarette per day) for the past year, and who meet other inclusion and exclusion criteria, are randomly assigned to receive self-help materials or self-help materials plus CM. Individuals in the CM group have the opportunity to win prizes, worth on average $1, $20, or $100, when they meet smoking abstinence criteria (CO < 8ppm and salivary cotinine < 10ng/mL). Participants meet with research staff 4 times/week during Weeks 1-4, 2 times/week during Weeks 5-8 and 1 time/week during Weeks 9-12. Follow-up interviews are scheduled 1, 3 and 6 months following the smoking quit date.

ELIGIBILITY:
Inclusion Criteria:

* meets diagnostic criteria for alcohol, cocaine or heroin abuse or dependence
* self-report daily smoking for at least the past year
* CO > 8ppm
* interested in quitting smoking while in treatment,
* minimum age 18 years old
* willing to provide names, addresses and phone numbers of individuals to assist in locating the patient for follow-up evaluations
* English speaking

Exclusion Criteria:

* current use of NRT
* current use of bupropion
* serious, uncontrolled psychiatric illness (e.g., acute schizophrenia, suicide risk)
* dementia (Mini-mental status score of <23)
* currently participating in another CM study at the clinic
* in recovery for pathological gambling

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Percent negative CO readings
Percent negative cotinine readings
Longest period of continuous abstinence

SECONDARY OUTCOMES:
Self-reported frequency and severity of smoking
Objective substance use
Self-reported substance use
Treatment retention

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M Alessi, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States